CLINICAL TRIAL: NCT00912496
Title: Phase I Randomized Study of the Safety, Dose Escalation, and Immunogenicity of Adjuvanted Influenza A/Anhui/05 Boosting in Subjects Previously Immunized With One or Two Doses of A/Vietnam/1203/04 or in Unprimed Individuals and Compared to Placebo
Brief Title: Booster Trial to 07-0019 With A/Anhui/05 With and Without MF59
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-0013; N01AI80003C
Record Dates: First submitted 2009-05-28; First posted 2009-06-03 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2011-10

CONDITIONS: Influenza
Keywords: Influenza, H5N1, vaccine, avian influenza
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Group 9: 2 dose prime (Experimental): Received two doses of A/Vietnam/1203/04 90mcg vaccine as prime (on Days 0, 28 in DMID 07-0019), will receive a booster dose of A/Anhui/05 vaccine (A) with or without MF59 adjuvant in DMID 08-0013 on Day 0.
  Interventions: Biological: MF-59; Biological: A/Anhui/05
- Group 8: 1 dose prime (Experimental): Received A/Vietnam/1203/04 90mcg vaccine as prime (Day 0 in DMID 07-0019), will receive a booster dose of A/Anhui/05 vaccine (A) with or without MF59 adjuvant in DMID 08-0013 on Day 0.
  Interventions: Biological: MF-59; Biological: A/Anhui/05
- Group 10: unprimed control/dose response group (Experimental): Unprimed control and dose response group of H5 vaccine naive volunteers will be added in DMID 08-0013 to receive two doses of A/Anhui/05 vaccine (A) with or without MF59 adjuvant or placebo on Day 0 and Day 28.
  Interventions: Biological: MF-59; Biological: A/Anhui/05; Drug: Placebo

INTERVENTIONS:
Biological: MF-59 — Doses of A/Anhui/05 vaccine (A) will be administered with or without MF59 adjuvant.
Biological: A/Anhui/05 — Monovalent inactivated surface antigen influenza A/H5N1 (modified Hemagglutinin and Neuraminidase of A/Anhui/01/2005) vaccine supplied in 5mL multi-dose vials with thimerosal [0.01%(w/v)] as a preservative. Each dose level includes both unadjuvanted and MF59C.1 adjuvanted formulations: 7.5, 15, 30, or 60 micrograms (mcg) of H5 Hemagglutinin per milliliter (mL) with MF59C.1, and 7.5, 15, 30, or 60 micrograms (mcg) of H5 Hemagglutinin per milliliter (mL) without MF59C.1 adjuvant.
Drug: Placebo — Sterile normal saline for injection (0.9% Sodium Chloride Injection, USP Preservative-Free).
  Arms: Group 10: unprimed control/dose response group

SUMMARY:
This research will study safety and the body's immune (defense system) responses, including anti-H5 flu antibodies (the body's protective proteins found in the blood), to an inactivated influenza "H5" bird flu, virus vaccine. Participants will be assigned by chance to receive the vaccine injections with and without an adjuvant, (substance that can improve vaccine effectiveness so less vaccine may be used) MF59, or placebo (inactive substance). Five different vaccine dose strengths will be evaluated. About 735 healthy participants, ages 18-49 will be asked to take part in this study. Study procedures include physical exam, blood sampling, and use of a memory aid. Volunteers will participate for up to 13 months.

DETAILED DESCRIPTION:
Severe disease in humans due to avian influenza viruses of the H5N1 subtype has raised considerable concern regarding the potential emergence of these viruses in pandemic form. Planning for control of such pandemics is of vital importance, and a cornerstone of this planning is the development of effective vaccines for H5N1. This study is designed to gather critical information on the safety, tolerability, and immunogenicity of booster vaccination with influenza A/Anhui/05 with and without the adjuvant MF59 in subjects previously primed with the clade 1 vaccine or unprimed individuals. Primary objectives are: to evaluate booster vaccination with a different variant/clade of A/Anhui/05 vaccine to assess possible prime for a broad immune response by 1 or 2 previous doses of A/Vietnam/1203/04; to compare 1-dose versus 2-dose priming of A/Vietnam/1203/04 followed by heterologous boosting with A/Anhui/05; to assess the safety of MF59 adjuvanted A/Anhui/05 vaccine in primed subjects; and to compare safety and immunogenicity of 1 and 2 doses of A/Anhui/05 with or without MF59 adjuvant, or to saline placebo, in a Phase I dose response study in naïve subjects. Up to 180 healthy adult subjects aged 18 through 49 (Subjects previously enrolled in 07-0019 will be eligible for 08-0013 even if they are older than 49 years of age at the time of enrollment into 08-0013.) who were previously enrolled in Division of Microbiology and Infectious Diseases (DMID) 07-0019 and received either 1 or 2 priming doses of A/Vietnam/1203/04 H5 influenza vaccine will be enrolled in this study. Additionally, approximately 555 healthy adult subjects aged 18 through 49 H5 vaccine naïve will be recruited to receive 2 doses, 28 days apart, of A/Anhui/05 vaccine with or without MF59 adjuvant or placebo. Entry criteria for the newly enrolled subjects will be the same as those used in DMID 07-0019. Because extensive safety data were collected for similar H5 vaccines, subjects will not be screened with clinical laboratory tests. The booster for Groups 8-9 will be randomized to 1 of 2 possible doses, with approximately 20 subjects per Group (allocation ratio 1:1) in each dose assignment: 3.75 micrograms (mcg) MF59, or 3.75 mcg. Newly enrolled, vaccine naïve subjects in Group 10 will be randomized to 1 of 9 possible dosages with or without MF59 adjuvant, with approximately 50 subjects in each dosage assignment: 3.75 mcg MF59, 3.75 mcg, 7.5 mcg MF59, 7.5 mcg, 15.0 mcg MF59, 15.0 mcg, 45.0 mcg MF59, 45.0 mcg, 90 mcg, or saline placebo with 3 groups of 35 subjects each, receiving different volumes of: one injection of 0.5 mL, one injection of 0.75 mL or 2 injections of 0.75 mL, for comparison. Volunteers will be observed in the clinic for at least 20 minutes after vaccination, and will maintain a Memory Aid to record oral temperature and systemic and local adverse events (AEs) and serious adverse events (SAEs) for 8 days after vaccination. Volunteers will be contacted by telephone 1 to 3 days after vaccination (approximately Day 2 post dose) to assess for the occurrence of AEs/SAEs, and they will return to the clinic 7 to 9 days after vaccination for AE/SAE and concomitant medication assessment, a targeted physical examination (if indicated), and review of the Memory Aid. Volunteers in Group 10 will return to clinic on Day 28 for review of eligibility criteria to receive Dose Number 2 of A/Anhui/05 or placebo. Volunteers in this group will then follow the same study schedule as following the first vaccination. All subjects will continue to be followed for 12 months after the last vaccination. It is anticipated that this study will enroll up to 735 subjects over 10-14 weeks. This

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 through 49 (Subjects previously enrolled in 07-0019 will be eligible for 08-0013 even if they are older than 49 years of age at the time of enrollment into 08-0013.) years old, who either were previously enrolled and received all scheduled vaccinations in Groups 8 and 9 under Division of Microbiology and Infectious Diseases (DMID) 07-0019, or are new subjects who deny exposure to H5 virus or participation in an H5 vaccine study.
* In good health, as determined by vital signs (heart rate <100 beats per minute (bpm); blood pressure: systolic less than or equal to 140 mm Hg and greater than or equal to 90 mm Hg; diastolic less than or equal to 90 mm Hg; oral temperature <100.0 degrees Fahrenheit), medical history to ensure stable medical condition and a targeted physical examination, as indicated, based on medical history. A stable medical condition is defined as no recent change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company, etc, or is done for financial reasons, as long as in the same class of medication, will not be considered a violation of the inclusion criterion. Any change to prescription medication due to improvement of a disease outcome will not be considered a violation of the inclusion criterion.
* Women of childbearing potential (not surgically sterile or postmenopausal for greater than or equal to 1 year) must not be pregnant as indicated by a negative pregnancy test (urine or serum) within 24 hours prior to vaccine administration.
* Women of childbearing potential who are at risk of becoming pregnant must have a history of practicing adequate contraception (i.e., barrier methods, abstinence, monogamous relationship with vasectomized partner, intrauterine devices, Depo-Provera, Norplant, oral contraceptives, contraceptive patches or other licensed, effective methods) in the 30 days prior to enrollment, and must agree to practice adequate contraception until 30 days following receipt of the last dose of vaccine.
* Able to understand and comply with planned study procedures.
* Able to provide informed consent prior to initiation of any study procedures and be available for all study visits.

Exclusion Criteria:

* Has occupational exposure to poultry, to include but is not limited to chicken, turkey, or duck farmer, factory worker in poultry processing plant, veterinary staff that handles poultry; has recreational exposure to poultry, e.g. raising poultry in 4-H club, duck hunter that slaughters/handles the "kill" or history of previous H5N1 vaccination or exposure (other than vaccination in Protocol 07-0019).
* Has a known allergy to egg proteins (egg or egg products), or other components of the vaccine (including thimerosal, polymyxin, neomycin, beta propiolactone, or nonylphenol ethoxylate).
* Is female of child-bearing potential who is breastfeeding or intends to become pregnant during the study period up to 30 days following receipt of the last dose of vaccine.
* Has immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematologic malignancy. An active neoplastic disease is defined as no neoplastic disease or treatment for neoplastic disease within the past 5 years.
* Has long-term use (greater than 2 weeks) of oral or parenteral steroids (glucocorticoids), or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
* Has a history of receiving immunoglobulin or other blood products within the 3 months prior to enrollment in this study.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study, or plans to receive any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) following each study vaccine.
* Has an acute or chronic medical condition that would render vaccination unsafe or would interfere with the evaluation of responses. This includes, but is not limited to: solicited reactogenicity symptoms, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients.
* Has a history of severe reactions following vaccination with contemporary influenza virus vaccines.
* Has an acute illness or has an oral temperature greater than 99.9 degrees Fahrenheit (37.7 degrees Celsius) within 3 days prior to enrollment.
* Has received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during the study period.
* Has any condition that would, in the opinion of the site principal investigator place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Has a diagnosis of schizophrenia, bipolar disease or other severe (disabling) chronic psychiatric diagnosis.
* Has been hospitalized for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Is receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, trifluopromazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensating are allowed enrollment into the study.
* Has known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* Has a history of alcohol or drug abuse in the 5 years prior to enrollment.
* Has a history of Guillain-Barré syndrome.
* Has any condition that the investigator believes may interfere with successful completion of the study.
* Plans to enroll in another clinical trial (that has a study intervention in the form of drug, biologic or device that could interfere with safety assessment of H5N1 vaccine) at any time during the study period.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 637 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titer, frequency of 4-fold or greater antibody titer increases, and proportion of subjects achieving a serum HAI antibody titer of 1:40 or greater against the 2 antigens being evaluated, A/Vietnam/1203/04 and A/Anhui/05 H5N1 virus. | 1 month and 6 months after last vaccination.
Local and systemic adverse event (AE) or serious adverse event (SAE) information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessments). | Duration of study.

SECONDARY OUTCOMES:
Geometric mean titer in primed versus unprimed subjects to A/Vietnam/1203/04 and A/Anhui/05. | Days 8 and 14 post-vaccination.
Geometric mean titer (GMT), frequency of 4-fold or greater increases and proportion of subjects achieving a titer of 1:40 or greater in neutralizing antibody titers against the two antigens being evaluated, A/Vietnam/1203/04 and A/Anhui/05 H5N1 virus. | 1 month and 6 months after last vaccination.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - Emory University School of Medicine - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - University of Iowa - Infectious Disease Clinic, Iowa City, Iowa
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Mayo Clinic, Rochester - Vaccine Research Group, Rochester, Minnesota
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke Translational Medicine Institute - Clinical Vaccine Unit, Durham, North Carolina
  - Vanderbilt University - Pediatric - Infectious Diseases, Nashville, Tennessee
  - University of Texas Medical Branch - Pediatrics - Infectious Diseases and Immunology - Galveston, Galveston, Texas
  - Group Health Research Institute - Seattle, Seattle, Washington